CLINICAL TRIAL: NCT01548391
Title: A Phase I Clinical Study Study of the Safety, Tolerability, and Pharmacokinetics of HX-1171 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biotoxtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012-0070
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
MeSH Terms: interventions — 1-O-hexyl-2,3,5-trimethylhydroquinone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- HX-1171 20 mg (20mg 1T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 40 mg (20mg 2T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 80 mg (20mg 4T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 160 mg (20mg 8T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 300 mg (200mg 1T, 20mg 5T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 600 mg (200mg 3T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 1200 mg (500mg 2T, 200mg 1T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 1500 mg (500mg 3T) (Experimental)
  Interventions: Drug: HX-1171
- HX-1171 2000 mg (500mg 4T) (Experimental)
  Interventions: Drug: HX-1171

INTERVENTIONS:
Drug: HX-1171 — 20mg, 200mg, 500mg

SUMMARY:
This study is designed to evaluate the safety, tolerability, and pharmacokinetics of HX-1171 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 40 years at screening.
* Be able to comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or gastrointestinal disorders.
* History of known hypersensitivity to drugs including HX-1171.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2012-03

PRIMARY OUTCOMES:
Safety (normal results for safety tests) | 14days
  Physical examination, Vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr